CLINICAL TRIAL: NCT05878262
Title: The Effect of Pre-emptive Analgesia on the Postoperative Pain in Children Undergoing Pediatric Stomatology Day Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaojing Li, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-IRB-183
Record Dates: First submitted 2023-05-09; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Ankyloglossia; Oral Mucoceles; Supernumerary Teeth
Keywords: pre-emptive analgesia; pediatric stomatology day surgeries; postoperative pain
MeSH Terms: conditions — Ankyloglossia; Tooth, Supernumerary; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The patients were randomly assigned into either the pre-emptive analgesia group or the control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient, parents, surgeon and pain assessor were all blinded to the study. Only investigator, anesthetist and the nurse delivering the analgesic to the child were not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-emptive analgesia group (Experimental): For the pre-emptive analgesia group children, the nurse delivered the ibuprofen suppository at the dose of 5-10 mg/Kg.
  Interventions: Drug: ibuprofen suppository
- control group (No Intervention): No medicine was taken for the control group.

INTERVENTIONS:
Drug: ibuprofen suppository — After the induction of anesthesia was performed, the nurse delivered the ibuprofen suppository at the dose of 5-10 mg/Kg for the pre-emptive analgesia group children.
  Other Names: no medicine
  Arms: pre-emptive analgesia group

SUMMARY:
The aim of this double-blinded, randomized, controlled trial was to test whether pre-emptive analgesia with ibuprofen suppository is effective for children undergoing pediatric stomatology day surgeries in the postoperative period.

DETAILED DESCRIPTION:
The recruited patients were randomly assigned into either the pre-emptive analgesia group or the control group. After the induction of anesthesia was performed, the nurse delivered the ibuprofen suppository at the dose of 5-10 mg/Kg for children of the pre-emptive analgesia group, and no measures were taken for the control group. All procedures of frenectomy, extraction of supernumerary teeth and excision of oral mucoceles were performed by a single surgeon. Postoperative pain was assessed using the Visual Analogue Scale (VAS), the Wong-Baker Faces Pain Rating Scale (WBS), and the Face, Leges, Activity, Cry, and Consolability (FLACC) scale, and Postoperative Parental Pain Assessment (PPPM) scale. The postoperative pain was measured 1, 4, and 24 hours after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* an age of 3-8 years; undergoing upper labial frenectomy, lingual frenectomy, extraction of supernumerary teeth, excision of oral mucoceles and the written informed consent from the parents or guardians.

Exclusion Criteria:

* children or parents refusal for study participation; intellectual disability, major systemic diseases; allergy to ibuprofen and other medications used in the study protocol.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The VAS scores for postoperative 1 hour pain | 1 hour after surgery
  The Visual Analogue Scale (VAS) is a line that is often 10 cm long with the markings "1"to"10","1"indicates no pain, and"10"represents very strong pain. The children were asked to mark a line on the scale to express the intensity of their pain at 1 hour postoperatively.
The WBS scores for postoperative 1 hour pain | 1 hour after surgery
  The Wong-Baker Faces Pain Rating Scale (WBS) contains six of faces from 0 point happy face representing no pain to 10 points crying face suggesting the strong pain. The children were asked to choose one face that indicating their state feelings at 1 hour postoperatively.
The FLACC scores for postoperative 1 hour pain | 1 hour after surgery
  The Face, Leges, Activity, Cry, and Consolability (FLACC) scale is an assessment tool that has five categories: facial expression, legs, activity, cry, and consolability. Each parameter is evaluated on a scale from 0 to 2, the total score is from 0-10 points. The FLACC scale was used by the researcher to assess pain at 1 hour after surgery.
The PPPM scores for postoperative 1 hour pain | 1 hour after surgery
  The Postoperative Parental Pain Assessment (PPPM) scale was is a valid and useful tool assessed by the parent or guardian for postoperative assessment of discharged children's pain. It has 15 items about children's emotional state, changes in appetite (eat less than usual , refuse to eat), behaviors, and activities, the total score is from 0-15 points. The PPPM scale was used by the parent or guardian to assess pain at 1 hour after surgery.
The VAS scores for postoperative 4 hours pain | 4 hours after surgery
  The Visual Analogue Scale (VAS) is a line that is often 10 cm long with the markings "1"to"10","1"indicates no pain, and"10"represents very strong pain. The children were asked to mark a line on the scale to express the intensity of their pain at 4 hours postoperatively.
The WBS scores for postoperative 4 hours pain | 4 hours after surgery
  The Wong-Baker Faces Pain Rating Scale (WBS) contains six of faces from 0 point happy face representing no pain to 10 points crying face suggesting the strong pain. The children were asked to choose one face that indicating their state feelings at 4 hours postoperatively.
The FLACC scores for postoperative 4 hours pain | 4 hours after surgery
  The Face, Leges, Activity, Cry, and Consolability (FLACC) scale is an assessment tool that has five categories: facial expression, legs, activity, cry, and consolability. Each parameter is evaluated on a scale from 0 to 2, the total score is from 0-10 points. The FLACC scale was used by the researcher to assess pain at 4 hours after surgery.
The PPPM scores for postoperative 4 hours pain | 4 hours after surgery
  The Postoperative Parental Pain Assessment (PPPM) scale was is a valid and useful tool assessed by the parent or guardian for postoperative assessment of discharged children's pain. It has 15 items about children's emotional state, changes in appetite (eat less than usual , refuse to eat), behaviors, and activities, the total score is from 0-15 points. The PPPM scale was used by the parent or guardian to assess pain at 4 hours after surgery.
The VAS scores for postoperative 24 hours pain | 24 hours after surgery
  The Visual Analogue Scale (VAS) is a line that is often 10 cm long with the markings "1"to"10","1"indicates no pain, and"10"represents very strong pain. The children were asked to mark a line on the scale to express the intensity of their pain at 24 hours postoperatively.
The WBS scores for postoperative 24 hours pain | 24 hours after surgery
  The Wong-Baker Faces Pain Rating Scale (WBS) contains six of faces from 0 point happy face representing no pain to 10 points crying face suggesting the strong pain. The children were asked to choose one face that indicating their state feelings at 24 hours postoperatively.
The FLACC scores for postoperative 24 hours pain | 24 hours after surgery
  The Face, Leges, Activity, Cry, and Consolability (FLACC) scale is an assessment tool that has five categories: facial expression, legs, activity, cry, and consolability. Each parameter is evaluated on a scale from 0 to 2, the total score is from 0-10 points. The FLACC scale was used by the researcher to assess pain at 24 hours after surgery.
The PPPM scores for postoperative 24 hours pain | 24 hours after surgery
  The Postoperative Parental Pain Assessment (PPPM) scale was is a valid and useful tool assessed by the parent or guardian for postoperative assessment of discharged children's pain. It has 15 items about children's emotional state, changes in appetite (eat less than usual , refuse to eat), behaviors, and activities, the total score is from 0-15 points. The PPPM scale was used by the parent or guardian to assess pain at 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fangqi Gong, doctor, Study Chair — Medical Ethics Committee, Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
After the raw research data are collected and collated, we will make the data including study protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code freely available to all researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data can be available now.
Access Criteria: researchers who study the pre-emptive analgesia, and pediatric stomatologists

REFERENCES:
- [Result] Zielinski J, Morawska-Kochman M, Dudek K, Czapla M, Zatonski T. The Effect of Pre-Emptive Analgesia on the Postoperative Pain in Pediatric Otolaryngology: A Randomized, Controlled Trial. J Clin Med. 2022 May 11;11(10):2713. doi: 10.3390/jcm11102713. PMID 35628840
- [Result] Kelly DJ, Ahmad M, Brull SJ. Preemptive analgesia II: recent advances and current trends. Can J Anaesth. 2001 Dec;48(11):1091-101. doi: 10.1007/BF03020375. PMID 11744585